CLINICAL TRIAL: NCT01178541
Title: Simultaneous Measurement of Both Fetal's Lateral Ventricles of the Brain
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: K111/2010
Record Dates: First submitted 2010-08-08; First posted 2010-08-10 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: ventricles; fetal; brain; asymmetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study designed to measure simultaneously the width of both lateral ventricles of the fetal brain. Thus, will enable to evaluate the normal asymmetry that may exist between the right and the left ventricles during the pregnancy.

DETAILED DESCRIPTION:
Study will enable to evaluate the normal asymmetry that may exist between the right and the left ventricles during the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* low risk pregnant women

Exclusion Criteria:

* high risk pregnant women

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: low risk pregnant women
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
width of lateral ventricles along the pregnancy | one year
  constructing a graph of the width of the lateral ventricles according to the gestational weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Vardimon, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Rotshild Women Health Center, Petah Tikva, Israel